CLINICAL TRIAL: NCT00931502
Title: Contemporary Treatment Of Stent Thrombosis In Acute Coronary Syndromes
Brief Title: Stent Thrombosis In Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: 214693; STR 001; 214693 (Other: UC Davis)
Record Dates: First submitted 2009-06-29; First posted 2009-07-02 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Stent Thrombosis; Acute Coronary Syndrome
Keywords: Stent thrombosis; Acute Coronary Syndrome; ACS; Stenting; Interventional Cardiology; Cardiology; Cardiovascular Research; Registry
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to better understand what treatment methods result in the best outcomes for patients who have heart attacks due to blood clots forming within stents.

DETAILED DESCRIPTION:
This is a multicenter registry that examines treatment strategies and outcomes in patients who present with acute coronary syndrome (ACS) due to stent thrombosis in the coronary arteries. This study will take place at potentially 8 medical centers throughout the State of California. A total of 800 patients will be enrolled into the registry, 100 patients from each of the eight participating California medical centers. UC Davis will serve as the core lab for this study.

Eligible subjects, patients who present to the hospital (medical center) with ACS due to stent thrombosis and receive a cardiac catheterization to treat the stent thrombosis, will be included in the retrospective analysis of this cardiac condition. Subjects who expire in hospital due to ACS with stent thrombosis will also be included in the retrospective analysis of this clinical registry. Patients, who consent for approval, will become eligible to participate in the 3-year prospective follow-up phase of the clinical registry. These patients will be followed for three years to learn more about long term clinical outcomes for this disease state.

There are no specific/special procedures required for this clinical registry. This is a registry for data collection only to correlate prescribed medical care with individual short- and long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age range will be ≥ 18 years old.
* Subjects will have an existing drug-eluting or bare metal stent.
* Subjects will have presented to the Medical Center with Acute Coronary Syndrome due to stent thrombosis as identified via cardiac catheterization.

Exclusion Criteria:

* Inability to consent/declined to participate in the prospective arm of the clinical registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had a heart attack or almost have had a heart attack due to blood clots forming within previously placed stents.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2008-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
To describe current real world practice in the treatment of ACS due to stent thrombosis. | 3 years

SECONDARY OUTCOMES:
To describe early and long term follow up of patients who are treated for ACS due to stent thrombosis. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Rogers, MD, Principal Investigator — University of California, Davis; Khung Keong Yeo, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Derived] Reeves RR, Patel M, Armstrong EJ, Sab S, Waldo SW, Yeo KK, Shunk KA, Low RI, Rogers JH, Mahmud E. Angiographic characteristics of definite stent thrombosis: role of thrombus grade, collaterals, epicardial coronary flow, and myocardial perfusion. Catheter Cardiovasc Interv. 2015 Jan 1;85(1):13-22. doi: 10.1002/ccd.25519. Epub 2014 May 7. PMID 24753053
- [Derived] Waldo SW, Armstrong EJ, Yeo KK, Patel M, Reeves R, Macgregor JS, Low RI, Mahmud E, Rogers JH, Shunk K. Procedural success and long-term outcomes of aspiration thrombectomy for the treatment of stent thrombosis. Catheter Cardiovasc Interv. 2013 Dec 1;82(7):1048-53. doi: 10.1002/ccd.25007. Epub 2013 Jul 2. PMID 23703925
- [Derived] Armstrong EJ, Yeo KK, Javed U, Mahmud E, Patel M, Shunk KA, MacGregor JS, Low RI, Rogers JH. Angiographic stent thrombosis at coronary bifurcations: short- and long-term prognosis. JACC Cardiovasc Interv. 2012 Jan;5(1):57-63. doi: 10.1016/j.jcin.2011.09.015. PMID 22230151